CLINICAL TRIAL: NCT04694469
Title: Comparison of Night-time and Daytime Operation on Outcomes of Supracondylar Humeral Fractures: A Prospective Observational Sudy
Brief Title: Comparison of Day-time and Night-time Operations of Supracondylar Humeral Fractures
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator M.D., Istanbul University
Other Study IDs: 2019/266
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Supracondylar Fracture; Morbidity
Keywords: supracondyler humerus fracture; night time operation; sleep deprivation; closed reduction and percutaneous pinning; CRPP
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Day: operated at 07:30 AM - 06:30 PM
  Interventions: Procedure: Closed reduction and percutaneous pinning (CRPP)
- Group Night: operated at 06:30 PM - 07:30 AM
  Interventions: Procedure: Closed reduction and percutaneous pinning (CRPP)

INTERVENTIONS:
Procedure: Closed reduction and percutaneous pinning (CRPP) — Operated for supracondylar humeral fractures

SUMMARY:
This study aims to investigate that performing supracondylar humerus fracture operations during daylight hours may have better results than performing them at night.

DETAILED DESCRIPTION:
Supracondylar humerus fractures are one of the most common traumatic fractures seen in children and their treatment usually requires immediate closed reduction and percutaneous pinning (CRPP). The presence of neurovascular complications associated with this fracture is considered an orthopedic emergency. For this reason, depending on the patient's operation time, the procedure should be performed at night under emergency conditions. Sleep deprivation, which is common in healthcare professionals, may affect patient safety due to disruptions in treatments and surgical procedures by reducing physician performance.

ELIGIBILITY:
Inclusion Criteria:

* aged 5 to 12 years
* had supracondylar humeral fractures,
* underwent CRPP
* under general anaesthesia
* American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

* Surgical procedures outside the operating room
* parental refusing the study protocol

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: paediatric population with supracondylar humeral fractures
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Morbidity | one month
  30 days morbidity
Operation duration | intraoperative
  time between anesthesia induction and anesthesia emergence

SECONDARY OUTCOMES:
Mortality | one month
  30 days mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet I. Buget, Assoc. Prof, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology; Nur Canbolat, MD, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology; Chasan Memet Chousein, MD, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Orthopedics and Traumatology; Ali Ersen, Assoc. Prof, Study Chair — Istanbul Unıversit Istanbul Faculty of Medicine, Orthopedics and Traumatology; Kemalettin Koltka, Assoc. Prof, Study Director — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology
Locations (1):
- Istanbul University, Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Tessler MJ, Charland L, Wang NN, Correa JA. The association of time of emergency surgery - day, evening or night - with postoperative 30-day hospital mortality. Anaesthesia. 2018 Nov;73(11):1368-1371. doi: 10.1111/anae.14329. Epub 2018 Aug 27. PMID 30151989
- [Background] Chacko AT, Ramirez MA, Ramappa AJ, Richardson LC, Appleton PT, Rodriguez EK. Does late night hip surgery affect outcome? J Trauma. 2011 Aug;71(2):447-53; discussion 453. doi: 10.1097/TA.0b013e3182231ad7. PMID 21825947